CLINICAL TRIAL: NCT06087432
Title: Investigation of the Effectiveness of Proprioceptive Neuromuscular Facilitation Exercises in Individuals With Temporomandibular Dysfunction With Forward Head Posture
Brief Title: Is PNF Application Effective on Temporomandibular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem ergezen, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-7705
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2023-11

CONDITIONS: TMD; TMJ Disorder; Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Rocabado's 6 x 6 exercise program has been found to be beneficial in reducing pain and increasing masticatory muscle function, as well as improving forward head posture, correcting limited joint mobility, muscle length limitation, and postural and functional limitations.
  Rocabado's 6x6 program includes 6 basic components: tongue rest position, TMJ rotation control, cervical spine release, shoulder girdle retraction and rhythmic stabilization technique. Rocabado's 6x6 exercises will be shown to both groups and 6 sets and 6 repetitions will be performed per day for 8 weeks
  Interventions: Other: Rocabado's 6x6 Exercises
- Group 2 (Experimental): Addition to Rocabado's, Proprioceptive neuromuscular facilitation (PNF) exercises will be applied to the neck and jaw with rhythmic stabilization (RS) and combined isotonic contraction (CIC) techniques.
  The patient will be placed supine on the treatment bed and asked to relax. The therapist's hands were placed according to PNF principles, depending on the applied technique and diagonality. Maximum resistance was provided to suit the needs of each individual First, the RS protocol will be applied and after a 2-minute rest interval, the exercise will continue with the KIK protocol applications. The expected duration of exercise exercises is 30 minutes. Maximum performance will be requested from the individual in all repetitions and the necessary verbal commands will be given for appropriate movement.
  Interventions: Other: Rocabado's 6x6 Exercises; Other: PNF Exercises

INTERVENTIONS:
Other: Rocabado's 6x6 Exercises — Rocabado's 6x6 program includes 6 basic components: tongue rest position, TMJ rotation control, cervical spine release, shoulder girdle retraction and rhythmic stabilization technique.
Other: PNF Exercises — Proprioceptive neuromuscular facilitation (PNF) exercises will be applied to the neck and jaw with rhythmic stabilization (RS) and combined isotonic contraction (CIC) techniques. The RS protocol consists of alternating isometric contractions for 10 seconds and does not involve movement. The KIK technique involves combined concentric, isometric and eccentric contraction of the agonist muscle without rest, with each contraction lasting 5 seconds. KIK exercises consist of 5-15 repetitions per set, depending on the individual's tolerance. Between sets, a 30-second rest will be included. First, the RS protocol will be applied and after a 2-minute rest interval, the exercise will continue with the KIK protocol applications. The expected duration of exercise exercises is 30 minutes. Maximum performance will be requested from the individual in all repetitions and the necessary verbal commands will be given for appropriate movement.
  Arms: Group 2

SUMMARY:
The goal of this clinical trial is to compare effects of Rocabado exercises which is conventional physiotherapy treatment alone vs. combine it with proprioceptive neuromuscular facilitation (PNF) in people with temporomandibular dysfunction (TMD) with forward head posture. The main question aims to answer:

- Does adding neck and jaw PNF techniques to the treatment affect the pain and functional status of the jaw compared to Rocabado exercises alone?

Participants will be randomized into two groups (Group 1: only Rocabado exercises, Group 2: Rocabado + PNF) and perform 8 weeks long exercises. They will be assessed in the beginning of the study and at the end of the 8th week.

DETAILED DESCRIPTION:
Infrared heat will be applied to the neck and face areas for 15 minutes for individuals with TMD with forward head posture in both groups. Then Group 1 will perform Rocabado exercises only, and Group 2 will perform PNF exercises in addition to Rocabado exercises. Exercises will be demonstrated and applied by a physiotherapist at the university clinic.

Pain intensity, pain threshold, TMJ functions, joint range of motion and Mandibular Function are among the parameters to be evaluated. All evaluations will be made by a blinded evaluator at baseline (baseline t=0), before exercise and after exercise (post-exercise, t=8.week).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of TMD according to the diagnostic criteria for temporomandibular disorders (RDC/TMD),
* Presence of trigger points in the relevant muscles,
* Presence of pain

Exclusion Criteria:

* Intra-articular or degenerative joint disorders and subluxation requiring urgent treatment;
* History of temporomandibular joint (TMJ) or cervical region surgery in the last 3 months;
* Treatment history from relevant areas;
* Presence of rheumatic diseases, including TMJ diseases;
* TMJ instability or fracture;
* Presence of perception-cognition disorder;
* Presence of chronic pain such as trigeminal neuralgia
* Orthopedic, neurological or rheumatological cervical disorders affecting jaw movements
* History of surgery in the jaw, head and neck area
* Presence of vertigo that prevents head movements during exercise

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Jaw Range of Motion (PMO) | 8 weeks
  Painless mouth opening (PMO) is a test in which the individual's maximum capacity to open her/his mouth without pain is measured in cm with a ruler.
Jaw Range of Motion (MMO) | 8 weeks
  Maximum mouth opening (MMO) is an outcome measure measured in cm in which the person opens their mouth to the maximum extent they can.
Jaw Range of Motion (MAMO) | 8 weeks
  Maximum assisted mouth opening (MAMO) is the maximum amount of opening that a person's mouth is forced to open with the help of the hand.
Pain Intensity | 8 weeks
  The person will be asked to mark the degree of pain he/she feels around the jaw on a ruler divided from 0 to 10 at equal intervals. According to VAS, 0 means "no pain" and 10 means "pain as bad as possible."

SECONDARY OUTCOMES:
Pressure Pain Threshold | 8 weeks
  Pressure pain threshold is measured by the physiotherapist with a hand algometer (TMD/RDC) in the examination form, including M. Temporalis (posterior, middle, anterior parts), M. Masseter (origo, body, insertion), posterior mandibular region and under the mandible, and M. sternocleidomastoideus and It will be measured on M. trapezius. The algometer will be applied vertically to the most painful point, increasing the pressure by 1kg/cm2 every three seconds until the patient feels pain, and the pressure value at which the pain begins will be recorded. 3 measurements will be made at 60-second intervals and the average value will be accepted as the pain threshold.
Functionality | 8 weeks
  The 8-item jaw functional limitation scale (JFLS-8) will be used to assess functionality. Each participant will be asked to report the level of restriction he or she has experienced for each of the eight items on the scale in the past month. Individuals will be told that the number "0" on the 10 cm horizontal line is no restriction and the number "10" is "severe restriction." Limitations in functionality will be determined by averaging each participant's responses.
Mandibular Functionality | 8 weeks
  The MFIQ is designed to assess the patient's perception of mandibular dysfunction. It consists of 17 items and a 5-point Likert scale is presented for each item. On this scale, the patient can indicate how much difficulty he or she has performing a particular mandibular movement or task. Likert scale scores; 0, no difficulty; 1, some difficulty; 3, very difficult; 4 means very difficult or impossible without help. The MFIQ also consists of a scoring range from 0 to 68. Here 0 indicates no mandibular dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen, PhD, Principal Investigator — Medipol University
Locations (1):
- Gizem Ergezen, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF